CLINICAL TRIAL: NCT01627821
Title: Evaluation of the Jarvik 2000 Left Ventricular Assist System With Post-Auricular Connector--Destination Therapy Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jarvik Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G100124
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jarvik 2000 Treatment (Active Comparator): Jarvik 2000 VAS, Post-Auricular Cable
  Interventions: Device: Jarvik 2000 VAS
- HeartMate II Control (Active Comparator): HeartMate II VAS Control
  Interventions: Device: HeartMate II

INTERVENTIONS:
Device: Jarvik 2000 VAS — Jarvik 2000 LVAD
  Arms: Jarvik 2000 Treatment
Device: HeartMate II — HeartMate II LVAD
  Other Names: HM II
  Arms: HeartMate II Control

SUMMARY:
This investigation will be conducted as an interventional intention-to-treat clinical study in a population of end stage heart failure patients who meet specific inclusion and exclusion criteria. The multi-center study will be prospective, dual-armed, non-blinded (open-label) and randomized, comparing a treatment group receiving the Jarvik 2000 LVAS with Post-Auricular Connector to an active control group treated with the PMA approved Thoratec HeartMate® II LVAS for Destination Therapy.

DETAILED DESCRIPTION:
Study Success for Primary Endpoint A will be established if the proportion of subjects in the Treatment Group meeting the Subject Success Criteria A, is determined to be non-inferior to that of the Control Group (at two years) according to the pre-specified statistical analysis.

Subject composite success requires the subject to achieve the Effectiveness Endpoint:

1. Two year actuarial survival
2. Freedom from procedures to repair, or replace the implanted device
3. Freedom from stroke resulting in a Modified Rankin Score of >3 at the two-year follow-up

Study Success for Primary Endpoint B will be established if the proportion of subjects in the Treatment Group meeting the Subject Success Criteria B is determined to be superior to that of the Control Group (at three years) according to the pre-specified statistical analysis.

Subject composite success requires the subject to achieve the Effectiveness Endpoint:

1. Three year survival
2. Freedom from the serious adverse event of drive cable or pump pocket infection

ELIGIBILITY:
Inclusion Criteria:

1. Cardiac transplantation ineligible.
2. Late stage heart failure in NYHA Class IIIb or IV for at least 45 of past 60 days.
3. Cardiac Index < 2.2 L / min / m2
4. LVEF = 25% or less
5. Patients on Optimal Medical Management (OMM) as defined in Section 9.2 OR dependent on intra-aortic balloon counter-pulsation for 7 days OR other temporary (indicated for 30 days use, or less) mechanical circulatory support for 7 days, OR supported with IV inotropes for 7 days and failing to respond.
6. BSA > 1.2 m2 and < 2.5 m2.

Exclusion Criteria:

1. History of cardiac transplantation or left ventricular reduction procedure.
2. Clinical conditions, other than heart failure, which could limit survival to less than three years.
3. Cause of heart failure due to, or associated with, uncorrected thyroid disease, obstructive / restrictive cardiomyopathy, pericardial disease, amyloidosis, dermatomyositis, or active myocarditis.
4. Intolerance to anti-coagulation or anti-aggregation therapy required for post-operative therapy.
5. Known sensitivity to products of bovine origin. The Jarvik 2000 incorporates a Hemashield vascular graft. Patients with a known sensitivity to products of bovine origin should not be implanted.
6. Chronic immunosuppression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2013-02; Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority to Control Group. | 2 years
  Study Success for Primary Endpoint A will be established if the proportion of subjects in the Treatment Group meeting the Subject Success Criteria A, is determined to be non-inferior to that of the Control Group (at two years) according to the pre-specified statistical analysis.
  Subject composite success requires the subject to achieve the Effectiveness Endpoint:
  1. Two year actuarial survival
  2. Freedom from procedures to repair, or replace the implanted device
  3. Freedom from stroke resulting in a Modified Rankin Score of >3 at the two-year follow-up

SECONDARY OUTCOMES:
Serious adverse events | 2 years
  Serious adverse events
Quality of life measures: Questionnaire | 2 years
  Kansas City Cardiomyopathy Questionnaire. There are 23 items. Scores from 0-100 in which a higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jarvik, MD, Study Chair — Jarvik Heart, Inc. SPONSOR
Locations (1):
- Columbia/NY Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No